CLINICAL TRIAL: NCT03389776
Title: Incidence of Postoperative Sore Throat in the Pediatric Population. An Observational Cohort Prospective Study
Brief Title: Postoperative Sore Throat in the Pediatric Population.
Acronym: POST
Status: Completed | Type: Observational
Sponsor: Istituto Giannina Gaslini (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nicola Disma, MD, Nicola Disma, MD, PhD, Istituto Giannina Gaslini
Other Study IDs: 2276
Record Dates: First submitted 2017-12-18; First posted 2018-01-04 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Anesthesia Morbidity; Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Anesthesia — Occurrence and severity of postoperative sore throat could be determined by various factors other than the pressure of the cuff alone. In particular, cuff pressure measurement, duration of anaesthesia, airway manipulations e.g. multiple insertion attempts, could all be factors determining the occurrence of postoperative sore throat.

SUMMARY:
Endotracheal tubes (ETT) and laryngeal mask airways (LMA) are devices used to help breathing whilst patients are asleep for surgery. Children may have a more satisfying experience if the rate of of post operative sore throat (POST) and hoarseness (PH) could be reduced. The incidence of POST and PH may be as high as 42% in children undergoing anesthesia. ETTs and LMAs require inflation of a cuff after insertion to obtain a seal to a patient's airway for them to be effective. It is recommended that cuff pressures are checked after insertion and inflation with a pressure checking device but this does not occur in all routine anesthetic practice. Overinflation of these cuffs may cause damage to the airway by exerting pressure on surrounding structures. Studies have shown both children and adults to have increased risk of POST with higher LMA pressure. The number of times it takes to successfully insert a LMA has also been associated with POST as has female gender and older age.

Similarly to LMAs, multiple insertion attempts of ETT insertion, female gender and a larger size are more likely to cause POST and PH.

Although patients with uncuffed have a higher incidence of POST than those with a cuffed ETT, when using cuffed tubes ETT, POST occurs more often as cuff pressure increases and should therefore be routinely measured.

The location of a patient's sore throat may vary. It may be intermittent or constant, or described as difficulty in swallowing, painful swallowing or hoarse voice and may there may be difference locations within the throat. In the current literature there is no one definition of what constitutes a sore throat or how or when it should be measured.

The hypothesis is that occurrence and severity of POST could be determined by various factors other than the pressure of the cuff alone. In particular, the pressure of cuff, the duration of anesthesia, the airway manipulations, could all be factors determining the occurrence of postoperative sore throat.

Based on the above hypothesis, Investigators planed to perform a prospective cohort study.

Aims: to determine the occurrence and severity of post-anaesthesia sore throat in children undergoing surgical procedures with LMA or ETT placement.

If clear factors are demonstrated for POST and PH in pediatric population then measures can be taken to reduce them and thereby improve outcome and patient satisfaction.

DETAILED DESCRIPTION:
The study is a prospective, descriptive study, involving patient interview and objective data collected as part of routine anesthetic care. No intervention will take place. Once identified from a theatre list, patients/parents will be approached preoperatively and consent taken to participate. If inclusion criteria are met and consent gained the preoperative questionnaire will be completed to obtain information regarding pain, nausea, sore throat, itching, thirst and hunger. Each symptom will be graded none, mild, moderate, severe. Intraoperative data will be collected after surgery whilst the child is in the recovery room. This is objective data obtained from the anesthetic chart. Prior to discharge to the ward the child will undergo a second interview answering the same questions as he/she did preoperatively (a further 1-2 minutes). Any child who has a sore throat in the recovery room will then be followed up 2 hours later on the ward with a further questionnaire. This will include questions about the location of the sore throat, severity and voice changes (5-10 mins). This will be the end of the participants input.

ELIGIBILITY:
Inclusion Criteria:

* Child age 5 or over
* General anaesthesia with LMA or ETT
* Children undergoing general, orthopaedic, urology, renal or plastic surgery

Exclusion Criteria:

* Other types of surgery
* Patients aged less than 5 years
* Patients affected by a significant cognitive delay
* Patients planned for anaesthesia with airway devices different from ETT and LMA

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A cohort of minimum 255 children will be prospectively collected from the elective surgical lists of Great Ormond Street Hospital, London, UK. Children 5 years of age or greater, scheduled for surgical procedures will be included.
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of sore throat | Six hours after anesthesia
  No pain, minimal pain, mild pain, severe pain

SECONDARY OUTCOMES:
Stridor | 6 hours after anesthesia
  Y/N
Laryngospasm | 6 hours after anesthesia
  Y/N
Oxygen desaturation | 6 hours after anesthesia
  Y/N
Time to oral intake | 6 hours after anesthesia
  Hours
Hospital discharge | 6 hours after anesthesia
  Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided